CLINICAL TRIAL: NCT02401945
Title: A Multicenter, Randomized, Open Label, Phase IIa Study Assessing the Efficacy, Safety and Duration of Effect of Intravitreal Injections of DE-120 as Monotherapy and With a Single Eylea® Injection in Subjects With Treatment-Naive Exudative Age-Related Macular Degeneration
Brief Title: A Safety and Efficacy Study of DE-120 Injectable Solution for Age-related Macular Degeneration
Acronym: VAPOR1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35-002
Record Dates: First submitted 2015-03-20; First posted 2015-03-30 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Age-Related Macular Degeneration
Keywords: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DE-120 Monotherapy (Experimental): DE-120 intravitreal injection given as monotherapy on a PRN basis
  Interventions: Drug: DE-120
- Eylea® and DE-120 Concomitant Therapy (Experimental): DE-120 intravitreal injection given on a PRN basis after Aflibercept (Eylea®) injection as an induction therapy.
  Interventions: Drug: DE-120; Drug: Aflibercept

INTERVENTIONS:
Drug: DE-120
Drug: Aflibercept
  Other Names: Eylea®
  Arms: Eylea® and DE-120 Concomitant Therapy

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of intravitreal (IVT) administration of DE-120 in subjects with treatment-naive active subfoveal choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* Provide signed written informed consent
* Diagnosis of active CNV secondary to wet AMD, with some subfoveal component in the study eye
* No evidence of subfoveal fibrosis or subfoveal RPE atrophy in the study eye
* At least one lesion in the study eye that meets minimal pathology criteria
* Best corrected visual acuity of 70 to 25 ETDRS letters in the study eye
* Best corrected visual acuity of 20/320 or better in the fellow eye
* Reasonably clear media and some fixation in the study eye

Exclusion Criteria:

Ocular

* Aphakic or has an anterior chamber intraocular lens in the study eye
* Received prior treatment with anti-VEGF, intravitreal corticosteroids or photodynamic therapy in the study eye
* Uncontrolled glaucoma despite anti-glaucoma therapy in the study eye
* Evidence of any ocular disease other than AMD in the study eye that may confound the outcome of the study
* History of vitrectomy in the study eye
* Need for ocular surgery in the study eye during the course of the trial
* Presence or history of certain ocular or periocular pathology or conditions that could limit ability to perform required study assessments in either eye and/or confound study results

Non-Ocular

* Allergy or hypersensitivity to study drug product, fluorescein dye or other study-related procedures and medications
* Current or history of certain systemic conditions, abnormalities or therapies that would render a subject a poor candidate for the study
* Participation in other investigational drug or device clinical trials within 30 days prior to randomization or planning to participate in other investigational drug or device clinical trials for the duration of the study
* Females who are pregnant or lactating and females of child-bearing potential who are not using adequate contraceptive precautions and men who do not agree to practice an acceptable method of contraception throughout the course of the study
* Unable to comply with study procedures or follow-up visits

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06-22 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in BCVA at Month 8 | Month 8

SECONDARY OUTCOMES:
Change from baseline in total lesion area at Month 8 | Month 8
Change from baseline in greatest linear dimension of the area of leakage at Month 8 | Month 8
Change in Central Subfield Thickness at Month 8 | Month 8

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Phoenix, Arizona
  - Bakersfield, California
  - Walnut Creek, California
  - Golden, Colorado
  - Altamonte Springs, Florida
  - Fort Myers, Florida
  - Indianapolis, Indiana
  - Portsmouth, New Hampshire
  - Charlotte, North Carolina
  - Dallas, Texas
  - Houston, Texas
  - McAllen, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah